CLINICAL TRIAL: NCT06901440
Title: Metabolic Biomarkers and Clinical Outcomes in Obesity: a Comparative Study of Surgical and Non-Surgical Cohorts
Brief Title: Bariatric Surgery for Obesity
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Elsayed Mohamed Abdallah, Internist at internal medicine department, faculty of medicine, Assiut University
Other Study IDs: NAssiutFs102030401989198932025
Record Dates: First submitted 2025-03-23; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Obesity and Obesity-related Medical Conditions; Bariatric Surgery Patients
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- -Intervention group: 25 adults (BMI ≥30) undergoing sleeve gastrectomy or Roux-en-Y gastric bypass.
- - Control group: 25 adults (BMI ≥30) managed with lifestyle/ dietary interventions.

SUMMARY:
Obesity has reached pandemic proportions worldwide, and its increased prevalence is associated with a plethora of metabolic disturbances. The obese state is characterized by increased adipose tissue mass and disturbed function resulting in systemic lipid spillover and low-grade inflammation, which may contribute to the development of comorbidities such as type 2 diabetes mellitus (T2DM) and cardiovascular disease. The crosstalk between various metabolic organs such as the gut, liver, adipose tissue, and skeletal muscle plays an important regulatory role in energy and substrate metabolism, which impacts metabolic health. The studies on the gut microbiota in host energy and substrate metabolism, & its relation to Obesity are neumerous, includes interventions that modify the gut microbiota composition and functionality with antibiotics , prebiotics & probiotics .

Obesity-associated with metabolic conditions such as ( Non alcoholic fatty liver diseases )NAFLD.

Obesity-associated NAFLD includes a spectrum of histological abnormalities ranging from steatosis to the inflammatory form of NAFLD, known as NASH. It is frequently seen in severe obesity, and its prevalence has been found to increase up to 90% in such patients in some countries.

So, in this study we compare liver status regarding degree of Steatosis among different patients, using Serum Biomarkers Scores and imaging techniques in obese patients undergo bariatric surgery ( case group ), and obese patients taking other lines of treatment ( Control group ); to detect if Bariatric surgery has better outcome for Steatosis and inflammatory markers than other lines of management for obesity.

- Research outcome measures:

a. Primary (main):

* Compare liver status regarding steatosis using Serum Biomarkers Scores in obese patients undergo bariatric surgery and obese patients taking other lines of treatment.
* Correlate these changes with weight loss and glycemic control.
* Secondary (subsidiary):
* Evaluate associations between these scores and insulin resistance, lipid profiles and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Two groups:

  * Intervention group: 25 adults (BMI ≥30) undergoing sleeve gastrectomy or Roux-en-Y gastric bypass.
  * Control group: 25 adults (BMI ≥30) managed with lifestyle/ dietary interventions.

Exclusion Criteria:

* Prior bariatric surgery, inflammatory bowel disease, antibiotic/probiotic use (past 3 months), or severe hepatic/renal dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese adults with (BMI ≥30) who has used any method of treatment for obesity
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Compare liver status regarding steatosis & Correlate changes with weight loss and glycemic control | one & half year
  Primary (main):
  * Compare liver status regarding steatosis using Serum Biomarkers Scores in obese patients undergo bariatric surgery and obese patients taking other lines of treatment.
  * Correlate these changes with weight loss and glycemic control

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided